CLINICAL TRIAL: NCT05532059
Title: A Phase Ⅱ, Open Label, Single-center Study of Lenvatinib and Tirelizumab Combined with Gemcitabine and Cisplatin (GPLET) in the Treatment of Advanced Cholangiocarcinoma
Brief Title: Lenvatinib, Tislelizumab Plus Gemcitabine and Cisplatin (GPLET) in Patients with Advanced Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220901
Record Dates: First submitted 2022-08-22; First posted 2022-09-08 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Advanced Cholangiocarcinoma
Keywords: Lenvatinib; Gemcitabine and Cisplatin; Tislelizumab; Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — lenvatinib; tislelizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- GPLET (Experimental): intravenous gemcitabine 1,000 mg/m2 and cisplatin 25 mg/m2 on days 1 and 8; oral lenvatinib 8 mg/day (<60kg) or 12 mg/ d（≥60kg）from days 1 to 21; intravenous tislelizumab 200 mg on day 15
  Interventions: Drug: Lenvatinib, tislelizumab, gemcitabine and cisplatin
- GP (Active Comparator): intravenous gemcitabine 1,000 mg/m2 and cisplatin 25 mg/m2 on days 1 and 8
  Interventions: Drug: gemcitabine and cisplatin

INTERVENTIONS:
Drug: Lenvatinib, tislelizumab, gemcitabine and cisplatin — Lenvatinib, tislelizumab, gemcitabine and cisplatin
  Arms: GPLET
Drug: gemcitabine and cisplatin — gemcitabine and cisplatin
  Arms: GP

SUMMARY:
Cholangiocarcinoma (CCA) is a heterogeneous group of cancers arising from the epithelial cells of bile ducts. Because of highly aggressive malignancy, most of the patients are diagnosed at an advanced stage and lose the chance to undergo surgery. As more effective and novel chemotherapy, targeted therapies, and immunotherapy become available, multiple treatments can be chosen for the patients with advanced CCA. Cytotoxic cell death during tumor chemotherapy triggers antigen release and induces strong anti-tumor effects of T cells. Tyrosine kinase inhibitors (TKI) can reduce the expression of PD-L1 and inhibit Treg cell infiltration, and together with immune checkpoint inhibitors, they can relieve tumor immunosuppressive microenvironment. Therefore,we aim to investigate the safety and efficacy of lenvatinib, tislelizumab combined with gemcitabine plus cisplatin (GPLET) in the treatment of advanced cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, unresectable advanced or metastatic cholangiocarcinoma patients.
* the world health organization (WHO)/ECOG physical state (PS) to 0 or 1.
* at least 1 RECIST 1.1 standard target lesions.
* not previously received immunotherapy, including but not limited to CTLA 4, PD-L1 or/and PD-1 inhibitors.
* adequate organ and bone marrow function, defined as follows: 9.0 g/dL or higher hemoglobin; neutrophil count 1.5 x 109 / L; platelet count 100 x 109 / L.

Exclusion Criteria:

* Active or previously documented autoimmune disease or inflammatory disease.
* Uncontrolled complications.
* History of other primary malignancies.
* Active infection.
* Women who are pregnant or breastfeeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
objective remission rate (ORR) | 4 cycle treatment (each cycle is 21 days)
  According to RECIST v1.1, the proportion of patients with at least one complete response (CR) or partial response (PR) (%)

SECONDARY OUTCOMES:
progression-free survival (PFS) | From date of randomization until the date of first documented progression, assessed up to 60 months
  The time between the date of randomization and the date of radiographic progression as defined by RECIST1.1
Overall survival time (OS) | From date of randomization until the date of death from any cause, assessed up to 60 months
  The time between the date of randomization and death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided